CLINICAL TRIAL: NCT06153966
Title: A Phase 1/2a Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intrathecally Administered ION717 in Patients With Prion Disease
Brief Title: PrProfile: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ION717
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION717-CS2; 2023-503355-98 (EudraCT Number)
Record Dates: First submitted 2023-11-21; First posted 2023-12-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Prion Disease
MeSH Terms: conditions — Prion Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ION717 + Placebo, Regimen 1 (Experimental): Participants will receive multiple doses of study drug (ION717 and placebo) during the 30-week double-blind treatment period; the order of doses is blinded. Participants will then receive multiple doses of ION717 during the 70-week open-label extension period.
  Interventions: Drug: ION717; Drug: Placebo
- ION717 + Placebo, Regimen 2 (Experimental): Participants will receive multiple doses of study drug (ION717 and placebo) during the 30-week double-blind treatment period; the order of doses is blinded. Participants will then receive multiple doses of ION717 during the 70-week open-label extension period.
  Interventions: Drug: ION717; Drug: Placebo

INTERVENTIONS:
Drug: ION717 — ION717 will be administered by IT injection.
Drug: Placebo — Placebo-matching ION717 will be administered by IT injection.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of intrathecal (IT) delivery of ION717.

DETAILED DESCRIPTION:
This is a first-in-human, randomized, multi-center study in participants with prion disease. Eligible participants will receive ION717 and placebo. The study will consist of a screening period of up to 6 weeks, a 30-week double-blind treatment period, a 70-week open-label extension period and a 32-week post-treatment period. During the double-blind period, the order of ION717 and placebo doses will be randomized and blinded to participants, study sites and the Sponsor. During the open-label extension period, all participants will receive ION717. Multiple dose levels will be tested.

ELIGIBILITY:
Key Inclusion Criteria

* A confirmed diagnosis of probable or definite prion disease.
* Early-stage prion disease at the time of Screening.
* Willing to meet all study requirements, including travel to Study Center, procedures, measurements and visits.
* Patients must have a caregiver who is ≥ 18 years old and who is able and willing to facilitate the patient's involvement, to the best of their ability, for the duration of the trial; caregivers must also be able and willing to provide information about themselves and the patient for the duration of the trial.
* Aged ≥ 18 at the time of informed consent.

Key Exclusion Criteria

* Clinically significant abnormalities in medical history, laboratory tests or physical examination that would render a patient unsuitable for inclusion.
* Any contraindication or unwillingness to undergo an MRI.
* Obstructive hydrocephalus, presence of a functional ventriculoperitoneal shunt for the drainage of cerebrospinal fluid (CSF) or an implanted central nervous system (CNS) catheter.
* Known brain or spinal disease that would interfere with the LP process, CSF circulation or safety assessment.
* Have any other condition, which, in the opinion of the Investigator would make the patient unsuitable for inclusion or could interfere with the patient participating in or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events. | Baseline up to Week 33

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ION717 | on Day 1 and Week 9
Area Under the Plasma Concentration-time Curve (AUC) of ION717 | on Day 1 and Week 9
Half-life (t1/2λz) of ION717 in Plasma | on Day 1 and Week 9
Cerebrospinal fluid (CSF) Concentration of ION717 | Pre-dose and at multiple points post-dose up to Week 33
Amount of ION717 Excreted in Urine | Post-dose on Day 1
Percent Change from Baseline in Prion Protein (PrP) Concentration in CSF | Pre-dose and at multiple points post-dose up to Week 33

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - UCLA Neurology Clinic, Los Angeles, California
  - University of Colorado Hospital, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Royal Melbourne Hospital, Parkville, Australia
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - McGill University Health Centre, Montreal, Quebec
- Hôpital Universitaire Pitié Salpêtrière, Paris, France
- University Medical Center Göttingen, Göttingen, Germany
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan, Italy
- Japan (3):
  - Mihara Memorial Hospital, Gunma, Isesaki-shi
  - National Center of Neurology and Psychiatry, Tokyo, Kodaira-shi
  - Neuromuscular Center Yoshimizu Hospital, Yamaguchi, Shimonoseki-shi
- Hospital Clinic De Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/